CLINICAL TRIAL: NCT05208398
Title: Apixaban in Patients With Left Ventricular Thrombus Post Myocardial Infarction; A Randomized Clinical Trial
Brief Title: Apixaban in Patients With Left Ventricular Thrombus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saud Al Babtain Cardiac Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2018-08
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Left Ventricular Thrombus
MeSH Terms: interventions — apixaban; Warfarin

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled clinical trial, two parallel active groups, with blinded primary study outcome assessor.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental): Apixaban, 5 mg oral tablets, on top of updated guidelines of acute coronary syndrome management recommendations
  Interventions: Drug: Apixaban
- Warfarin (Active Comparator): Warfarin, oral tablets, to achieve international normalized ratio (INR) of 2-3, on top of standards of care, as per updated guidelines of acute coronary syndrome management recommendations
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — 5 mg twice daily, on top of standards of care.
  Other Names: Eliquis
  Arms: Apixaban
Drug: Warfarin — Warfarin, oral tablets, to achieve international normalized ratio (INR) of 2-3, on top of standards of care, as per updated guidelines of acue coronary syndrome management recommendations
  Arms: Warfarin

SUMMARY:
Open label randomized controlled clinical trial to evaluate the efficacy and safety of apixaban versus warfarin in treating left ventricular thrombus in patients with acute or recent myocardial infarction (MI).

ELIGIBILITY:
Inclusion Criteria:

All the following criteria must be fulfilled:

* Ages between 18 and 80 years,
* History of anterior wall MI, either acute (within a week) or recent (within a month)
* Evident left ventricular thrombus (LVT) by transthoracic echocardiography,
* Naïve to oral anticoagulants (OAC)
* stable to start OAC

Exclusion Criteria:

* Other indications for OAC,
* Patients with contraindications for OAC,
* Right ventricular thrombus or atrial thrombus,
* History of confirmed stroke or other systemic embolization within the previous six months,
* High bleeding risk,
* Severe renal impairment,
* Patients with expected difficulties to follow the INR strictly.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Resolution of left ventricular thrombus | 3 months
  Transthoracic, noncontrast, echocardiographic assessment.

SECONDARY OUTCOMES:
Resolution of left ventricular thrombus | 6 months
  Transthoracic, noncontrast, echocardiographic assessment.
Safety outcome | 3-6 months
  Major Adverse Cardiovascular Events (MACE) or any relevant bleeding according to the Bleeding Academic Research Consortium (BARC) classification

CONTACTS AND LOCATIONS:
Locations (1):
- Saud AlBabtain Cardiac Center, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
No plan to share.